CLINICAL TRIAL: NCT03807167
Title: Apathy in Late Life Depression: New Biomarkers Using Actimetry and Magnetic Resonance Imaging
Acronym: ACTIDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC18_8833_ACTIDEP
Record Dates: First submitted 2018-12-07; First posted 2019-01-16 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental)
  Interventions: Other: Mattis Dementia Rating Scale; Other: Unified Parkinson 's Disease Rating Scale-III; Other: Mini Neuropsychiatric Investigation; Other: Montgomery and Asberg depression Rating Scale; Other: Clinical Global Impression; Other: Apathy diagnostic criteria; Other: walking speed test; Other: accelerometer presentation; Other: data acquisition from the accelerometer; Other: Apathy Evaluation Scale,; Other: fatigue Visual Analog Scale; Other: executive function; Other: MRI; Other: Apathy Motivation Index
- healthy controls (Active Comparator)
  Interventions: Other: Mini Neuropsychiatric Investigation; Other: Montgomery and Asberg depression Rating Scale; Other: Clinical Global Impression; Other: accelerometer presentation; Other: data acquisition from the accelerometer; Other: executive function; Other: MRI

INTERVENTIONS:
Other: Mattis Dementia Rating Scale — This scale was developed to assess the cognitive status of patients with neurodegenerative diseases. There are 37 items that are presented in a fixed order and grouped into five sub-scales: attention, initiation, construction, conceptualization and memory. Patients and healthy subjects with a score below 125 are not included because of major cognitive impairment.
  Arms: Patients
Other: Unified Parkinson 's Disease Rating Scale-III — This scale is used to rate the severity of extra-pyramidal symptoms (akinesia, rigidity and tremors). These symptoms may be the cause of reduction of motor activity apart from any reduction in motivation, they onstitute a confounding factor that it should be controlled.
  Arms: Patients
Other: Mini Neuropsychiatric Investigation — This is a structured interview that allows rapid screening in about 20 minutes of troubles Psychiatric. It is based on short questions to which the patient must answer yes or no and on a decision tree. Patients must validate clinical diagnoses of depression.
Other: Montgomery and Asberg depression Rating Scale — This scale is composed of 10 items from 0 to 6 from a semi-structured interview, to obtain a total depression score of 0 to 60 (0 no depression, 60 maximum intensity of depression).
Other: Clinical Global Impression — heterosexual assessment that rates the severity of symptoms suicidal and changes in suicidal symptoms. Any subject with a score greater than 4 is not included.
Other: Apathy diagnostic criteria — The clinical criteria make it possible to make a diagnosis of apathy with a functional repercussion. It is based on a lack of motivation felt by the patient, causing a functional or social impact that is not the consequence of a disturbance of consciousness or a disability engine. The cognitive, emotional and behavioral dimensions are affected.
  Arms: Patients
Other: walking speed test — The patient is timed to walk 10m. A speed <1m / sec is a criterion exclusion because it shows severe sarcopenia and constitutes a bias.
  Arms: Patients
Other: accelerometer presentation — accelerometer presentation and pose
Other: data acquisition from the accelerometer — withdrawal of the accelerometer and data acquisition from the accelerometer
Other: Apathy Evaluation Scale, — clinician version and near-helping version. It's a hetero rating scale from an interview semi structured by a trained clinician. It assesses cognitive, emotional and behavioral apathy than three items of various apathy. The total score ranges from 18 (total absence of apathy) to 72.
  Arms: Patients
Other: fatigue Visual Analog Scale — To date, there is no valid fatigue scale in the depression of the elderly subject, a fortiori in French. The fatigue scale in adult depression includes has been validated with an EVA (Visual Analogue Scale) (38). We therefore propose to use this type of evaluation to control this aspect.
  Arms: Patients
Other: executive function — * Modified Card Sorting Test MCST(Modified Card Sorting Test) (Wisconsin Test): This test assesses conceptualization, attention and mental flexibility using a deck of cards.
  * Trail Making Test (TMT): This test is used to assess mental flexibility.
  * Fluences verbal: This test tests the capacities of setting up search strategies in memory semantics and oral language.
  * Stroop Paradigm: This test is used to evaluate the resistance to interference, ie the patient's ability to inhibit some over-learned and automated responses.
Other: MRI — An MRI lasting 30 minutes is programmed
Other: Apathy Motivation Index — This is a self-questionnaire of 18 items, each side on a 5-level Likert scale (0: not everything at 4: very often). It differentiates between "behavioral" apathy and "social" apathy.
  "Emotional".
  Arms: Patients

SUMMARY:
Old age (> 60 years) is at high risk to develop major depression disorders (MDD). MDD doubles the risk for subsequent cognitive disorders and dementia. Apathy (i.e. the lack of motivation) is a core problem in depression in older age and is frequently associated with cognitive decline in people who have mild cognitive disorders. The investigator propose here to combine actimetry (the measurement of motor activity using a simple device worn at the wrist) and brain imaging to show that it's possible to measure apathy using actimetry in a population of elders with MDD. Having shown that apathy can reliably be measured with actimetry and that it is associated with brain abnormalities, the investigator will be able to test whether actimetry can predict cognitive decline in elders with MDD and can be routinely used in a day-to-day medical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* 60 years and above
* Major depressive disorder (either late-onset or early onset)
* Ambulatory settings
* Both uni and bipolar depression will be considered Healthy controls
* 60 years and above
* No psychiatric disorders, including no major depressive disorder
* No non-inclusion criteria

Exclusion Criteria:

* Patients and healthy controls
* Major cognitive disorders (< 125 on the Mattis dementia rating scale and a major cognitive disorders diagnostic according to the DSM5 (Diagnostic and Statistical Manual of Mental Disorders) criteria).
* Other neurological conditions (stroke, Parkinson's disease and seizures), severe and inflammatory disorders (ex: severe arthroses which limits movements, spondylarthritis)
* Severe sarcopenia: speed walk < 1 meter/second
* Extrapyramidal syndrome
* High suicidal risk
* Anti-psychotic prescription
* Participant who are unable to provide clear consent, under legal protection
* MRI contra-indication

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Actimetry | 3 days
  Measure of actimetry: immobility, transfer, walking, movement given by the accelerometer

SECONDARY OUTCOMES:
grey matter density | at Day 3 (+/- 2 days)
  Magnetic Resonance Imaging brain metrics: grey matter density
cortical thickness | at Day 3 (+/- 2 days)
  Magnetic Resonance Imaging brain metrics: cortical thickness;
diffusion tensor imaging, | at Day 3 (+/- 2 days)
  Magnetic Resonance Imaging brain metrics: diffusion tensor imaging,
Rest functional connectivity analysis | at Day 3 (+/- 2 days)
  Magnetic Resonance Imaging brain metrics: regional cerebral blood flow
pulsatility. | at Day 3 (+/- 2 days)
  Magnetic Resonance Imaging brain metrics: pulsatility.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre Mémoire de Ressources et de Recherche (CMRR),, Nice
  - CHU Pontchaillou, Département de Radiologie et d'Imagerie Médicale, Rennes
  - Centre Hospitalier Guillaume Régnier, Pôle Hospitalo-Universitaire de Psychiatrie Adulte, Rennes
  - CHU Bretonneau, Consultations Intersectorielles de Gérontopsychiatrie, Tours
  - CHU Bretonneau,CIC, Tours
  - Service de Radiologie- Neuroradiologie,CHU bretonneau, Tours